CLINICAL TRIAL: NCT02471742
Title: Nipple Areolar-complex Sparing Mastectomy After Neo-adjuvant Chemotherapy: Evaluation of Local Oncologic Safety in a Cohort Study Analysis
Brief Title: NAC Sparing Mastectomy After Neo-adjuvant Chemotherapy
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: INT 177/13
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- NAC-PC: patients treated with neoadjuvant chemotherapy and NAC-sparing mastectomy
  Interventions: Procedure: NAC-sparing mastectomy
- NAC: patients treated NAC-sparing mastectomy and adjuvant therapy
  Interventions: Procedure: NAC-sparing mastectomy
- PC: patients treated with neoadjuvant chemotherapy and conventional mastectomy
  Interventions: Procedure: conventional mastectomy

INTERVENTIONS:
Procedure: NAC-sparing mastectomy — patients treated with mastectomy with conservation of nipple-areola complex
  Groups: NAC; NAC-PC
Procedure: conventional mastectomy — patients treated with mastectomy without conservation of nipple-areola complex
  Groups: PC

SUMMARY:
Nipple areolar-complex (NAC) sparing mastectomy, extending the concept of skin-sparing mastectomy, allows to leave the nipple-areola complex intact and to provide a better cosmetic result. Large operable T2-T3 breast cancer (BC), treated with neoadjuvant chemotherapy, may theoretically appear suitable for this surgical option, alternative to conventional mastectomy or breast conserving surgery in case of unfavorable size of the breast, when a good response to neoadjuvant chemotherapy has been achieved.

DETAILED DESCRIPTION:
From January 2009 to May 2013, 422 BC patients were progressively accrued to NAC-sparing mastectomy, of which 361 invasive BC patients underwent NAC-sparing mastectomy as first treatment (NAC-group), whereas 61 T2-T3 invasive BC patients underwent surgery after primary chemotherapy (NAC-PC group). 151 BC patients underwent primary chemotherapy and conventional mastectomy (PC group) from 2004 to 2009, has been evaluated as comparative group respect to NAC-PC group.

Using propensity score matching, local disease-free survival (LDFS) in NAC-PC patients was first compared with that in PC patients.

The NAC-PC cohort was then compared to NAC patients in terms of LDFS using two different matching criteria, one with tumor size after neoadjuvant chemotherapy and one with tumor size before neoadjuvant chemotherapy as balancing covariates.

ELIGIBILITY:
Inclusion Criteria:

T2-T3 N0-N1 breast cancer (NAC-PC and PC groups). T1-T3 N0-1 M0 breast cancer (NAC-group) In our series of NAC-sparing mastectomy patients, with or without treatment with neo-adjuvant chemotherapy, the selection of patients for NAC-sparing mastectomy has been made on the basis of the following criterions: tumor nodule without adherence to the skin, no nipple retraction, retroareolar main duct free for neoplastic tissue inside at frozen section examination. Furthermore, patients were considered still eligible for NAC-sparing mastectomy even if the tumor lies in close proximity (<1 cm) to the NAC at physical and radiological examination.

Exclusion Criteria:

(NAC-PC and PC groups). Exclusion criteria for the present study were all the other breast cancer patients, particularly T4 breast cancer with inflammatory or ulcerated breast cancer before chemotherapy and patients with synchronous distant metastases. Patients affected with other clinical diseases (i.e. cardiovascular diseases) conditioning the optimal therapeutic strategy were excluded.

For NAC-sparing mastectomy, exclusion criterions were nipple retraction, Paget's disease, inflammatory changes of the breast and bloody discharge from the nipple. The study did not exclude women with prior breast augmentation, heavy smokers, obese patients.

-

Ages: 23 Years to 77 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both the population of patients treated with neoadjuvant chemotherapy (NAC-PC and PC groups) were T2-T3 N0-N1 breast cancer.
  The population of patients who underwent NAC-sparing mastectomy as primary therapy (NAC-group) were T1-T3 N0-1 M0 breast cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 573 (Actual)
Dates: Start 2004-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
local disease free survival | 11 years
  this study evaluates the local safety of NAC-sparing mastectomy compared with conventional mastectomy after neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Agresti, MD, Principal Investigator — Istituto Tumori Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, MI, Italy